CLINICAL TRIAL: NCT01089075
Title: Phase IV Study to Evaluate the Neuropsychological Effects of Hydrocortisone Substitution in Patients With Partial Adrenal Insufficiency After Traumatic Brain Injury or Subarachnoidal Haemorrhage
Brief Title: Neuropsychological Effects of Hydrocortisone in Patients With Partial Adrenal Insufficiency
Acronym: CSMünchen01
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment of suitable patients.
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-014909-14
Record Dates: First submitted 2010-02-02; First posted 2010-03-18 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Partial Corticotrope Insufficiency
Keywords: neuropsychological effects of hydrocortisone replacement
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo/20 mg hydrocortisone (Placebo Comparator): Order of study treatment: 7 days placebo followed by 7 days 20 mg hydrocortisone
  Interventions: Drug: Hydrocortisone; Drug: Placebo
- 20 mg hydrocortisone/placebo (Active Comparator): Order of study treatment: 7 days 20 mg hydrocortisone followed by 7 days placebo
  Interventions: Drug: Hydrocortisone; Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — 20 mg po for 7 days (2 tablets)
  Other Names: Hydrocortison GALEN 20 mg
Drug: Placebo — 2 tablets po
  Other Names: P-Tabletten 7 mm Lichtenstein

SUMMARY:
The purpose of this study is to evaluate the efficacy of hydrocortisone replacement therapy in patients with partial cortisol deficiency after traumatic brain injury or subarachnoid hemorrhage on cognitive function.

DETAILED DESCRIPTION:
This is a controlled, randomized, double-blind, placebo-controlled, crossover, interventional study. The benefit of replacement in partial corticotropic failure on brain function (cognition), especially in cases with borderline low cortisol levels after stimulation is unknown.

Moreover, since glucocorticoids might affect hGH secretion, the effect of hydrocortisone on hGH secretion reflected by IGF-1 levels will be assessed. If IGF-1 is below 2 SD at the end of the study, hGH secretion will additionally be determined by a GHRH-arginine-test.

An improved cognition in TBI and SAH patients with partial corticotropic insufficiency would give a new treatment option in this population which may lead to better quality of life and an enhanced rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (male and female) between 18 and 75 years
* 1 -12 month after TBI or SAH before prescreening
* Cortisol level 100-180 ng/ml after stimulation with ACTH
* Written informed consent by patient or a legally accepted representative

Exclusion Criteria:

* Pregnancy and lactation period (during study treatment)
* Concomitant or previous high-dose therapy with glucocorticoids; previous treatment with glucocorticoids will be accepted, if it has been low dose (i.e. lower than the Cushing threshold) and has been stopped at least 3 months before study participation
* Suspected or known hypersensitivity to hydrocortisone or any of its components
* Albumine less than 2,5 g/dl
* Suspected or known drug or alcohol abuse
* Planned treatment for thyroid dysfunction or a planned change in established thyroid treatment
* Any condition which in the opinion of the investigator makes the patient unsuitable for inclusion.
* Participation in another clinical trial with investigational new drugs
* Severe medical or psychiatric disease
* Change of dosage of any other drug which might influence the corticotrope axis or cognitive function (e.g. antidepressive treatment) during the last 3 weeks
* Oral contraceptives
* Severe disturbances in articulation, visual faculty or hearing
* Any elective surgery or medical treatment planned in the observation period
* Intensive Care treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes in score of alertness test (TAP)- interindividual differences | day -5 to - 0 (before start of study treatment), day 7 (after 7 days treatment with Hydrocortisone or Placebo, day 14 (after 7 days treatment with Hydrocortisone or Placebo)

SECONDARY OUTCOMES:
Changes in score of Alertness Test (TAP) - intraindividual differences | day -5 to - 0 (before start of study treatment), day 7 (after 7 days treatment with Hydrocortisone or Placebo, day 14 (after 7 days treatment with Hydrocortisone or Placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Günter K. Stalla, Prof. Dr., Study Director — Max-Planck-Institute, Munich
Locations (1):
- Schön Klinik Bad Aibling, Bad Aibling, Bavaria, Germany

REFERENCES:
- See also: Click here for more information about endocrinological diseases — http://www.endokrinologie.net/dge.php